CLINICAL TRIAL: NCT01970527
Title: RADVAX: A Stratified Phase II Dose Escalation Trial of Stereotactic Body Radiotherapy Followed by Ipilimumab in Metastatic Melanoma
Brief Title: Phase II Trial of Stereotactic Body Radiotherapy Followed by Ipilimumab in Treating Patients With Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in standard of care
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9031; NCI-2013-01757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9031 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (stereotactic body radiotherapy, ipilimumab) (Experimental): Patients undergo a total of 3 fractions of stereotactic body radiotherapy between days 1-13. Patients then receive ipilimumab IV every 3 weeks. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT

SUMMARY:
This phase II trial studies how well stereotactic body radiotherapy and ipilimumab work in treating patients with stage IV melanoma. Stereotactic body radiotherapy (SBRT) may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Monoclonal antibodies, such as ipilimumab, target certain cells to interfere with the ability of tumor cells to grow and spread. Giving SBRT with ipilimumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility and immune-related clinical responses associated with SBRT when given in conjunction with ipilimumab.

SECONDARY OBJECTIVES:

I. To determine late toxicity and immune pharmacodynamic changes after SBRT followed by ipilimumab.

OUTLINE:

Patients undergo a total of 3 fractions of stereotactic body radiotherapy between days 1-13. Patients then receive ipilimumab intravenously (IV) every 3 weeks. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 60 days, and then every effort will be made to obtain records of patients during this follow up, and permission will be sought for the investigators and/or study team to re-contact the patient directly with regard to health status and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Previously treated or previously untreated stage IV melanoma by American Joint Committee on Cancer (AJCC) staging criteria
* Presence of an index lesion between 1 and 5 cm
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Signed informed consent document
* Adequate renal, hepatic, and hematologic indices for ipilimumab therapy
* Ability to tolerate stereotactic body radiation therapy (e.g. lie flat and hold position for treatment)

Exclusion Criteria:

* Prior systemic therapy within 14 days of study enrollment; patients must be adequately recovered from prior systemic therapy side effects as deemed by the treating investigator
* Clinical contraindication to stereotactic body radiotherapy (e.g. active systemic sclerosis, active inflammatory bowel disease if bowel is within target field, etc)
* Presence of central nervous system metastasis (including active brain metastasis); active brain metastasis would be defined as untreated brain metastases; if the brain metastases have received prior treatment (usually either with surgery or radiation), they are no longer active
* Long-term use of systemic corticosteroids; patients with replacement steroids and not immunosuppressive steroids may enroll in the study
* Prior radiation therapy (RT) that precludes the delivery of SBRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2018-11-03 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Rengan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of January 2018, 23 participants consented to the study during accrual duration of 36 months. The participants with metastatic melanoma were recruited from the clinic at Department of Radiation Oncology, University of Washington Medical Center.
Pre-assignment Details: The total number of participants that consented to the study are 23, however 1 participant was a screen-fail due to brain metastasis.
Groups:
- Bone or Lung Index Lesion: Participants with bone or lung index lesion with prescription dose per fraction to the Planning Target Volume (PTV) of 8 Gy per fraction. The total dose for dose level 1 (our starting dose level) will be 24 Gy over 3 fractions. If we encounter a dose limiting toxicity, we will then reduce our total dose to dose level -1. The total dose for dose level -1 will be 12 Gy over 2 fractions.
- Liver or Subcutaneous Index Lesion: Participants with liver or subcutaneous index lesion with prescription dose per fraction to the Planning Target Volume (PTV) of 6 Gy per fraction. The total dose for dose level 1 (our starting dose level) will be 18 Gy over 3 fractions. If we encounter a dose limiting toxicity, we will then reduce our total dose to dose level -1. The total dose for dose level -1 will be 12 Gy over 2 fractions.
Period: Pre-treatment/Baseline
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion
Started | 9 | 14
Completed | 8 | 14
Not Completed | 1 | 0
Not completed — Screen fail- participant had brain mets | 1 | 0
Period: Treatment
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion
Started | 8 | 14
Completed | 8 | 11
Not Completed | 0 | 3
Not completed — Disease progression | 0 | 1
Not completed — Participant did not tolerate Ipilimumab | 0 | 1
Not completed — Death | 0 | 1
Period: Follow-up Clinic Visit
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion
Started | 8 | 11
Completed | 7 | 8
Not Completed | 1 | 3
Not completed — Disease progression | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 14 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Clinical Response, Defined as Proportion of Patients Treated at the Maximum-tolerated Dose (MTD) Who Achieve Either a Complete or Partial Immune-related Response
Description: Scored on a non-index lesion using immune-related response criteria according to immune-related Response Evaluation Criteria in Solid Tumors version 1.1. The number of immune-related responses will be tabled by stratum and SBRT fraction dose level. At the MTD, the immune-related response rate and 95% exact confidence interval will be estimated separately for previously untreated and previously treated metastatic patients.
Time Frame: Up to 60 days after last ipilimumab injection
Population: Arms were stratified during tx for safety reasons, but the stated objective to calculate response rate per strata was re-assessed. Due to low accrual per-strata calculations lack the statistical power to draw robust conclusions. Results were not stratified during the statistical analysis of the study data and are reported as such here.
Measure: Count of Participants; unit: Participants
Groups:
- Stable Disease: Patients with Stable disease at any point in follow up
Arm/Group | Stable Disease
Number analyzed (Participants) | 22
Participants | 6

2. Primary Outcome: Immune-related Progression-free Survival (irPFS)
Description: irPFS will be estimated by the Kaplan-Meier method separately for previously untreated and previously treated metastatic patients who were treated at the MTD..
  For some patients no scans were available for irRECIST reads, in which case change of management was determined to be the point of progression.
Time Frame: Time from first day of radiotherapy to first documented immune-related progressive disease, death due to any cause or last patient contact alive and progression-free, assessed at 6 months
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Days
Groups:
- Immune Naive: Previously untreated metastatic melanoma patients
- Immune Resistant: Previously treated metastatic melanoma patients
Arm/Group | Immune Naive | Immune Resistant
Number analyzed (Participants) | 15 | 6
Days | 131 (30.4) | 121 (50.3)
Statistical Analysis 1: Comparison: Immune Naive vs Immune Resistant; Test type: Superiority; p = 0.67, Log Rank

3. Primary Outcome: Late Toxicities, Graded According to the Radiation Therapy Oncology Group/European Organization for Research, the Treatment of Cancer Late Morbidity Scoring System, and the Common Terminology Criteria for Adverse Events Version 4.0
Description: Defined generally as an adverse event associated with the treatment which occurs beyond 30 days after last injection (i.e., adverse events which are observed months after treatment are most likely associated with SBRT). All dose-limiting toxicities and late toxicities will be graded and tabled by lesion site stratum and SBRT fraction dose level. Toxicity attribution to either SBRT or ipilimumab will be described if possible.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion
Number analyzed (Participants) | 8 | 14
Participants | 2 | 1

4. Primary Outcome: Overall Survival
Description: Will be estimated by the Kaplan-Meier method separately for previously untreated and previously treated metastatic patients who were treated at the MTD.
Time Frame: Time from first day of radiotherapy to death due to any cause or last patient contact alive, assessed at 12 months
Population: Arms were stratified during tx for safety reasons, but the stated objective to calculate response rate per strata was re-assessed. Due to low accrual per-strata calculations lack the statistical power to draw robust conclusions. Results were not stratified during the statistical analysis of the study data and are reported.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Immune Naive | Immune Resistant
Number analyzed (Participants) | 16 | 6
Days | 154 (327.6) | 307.5 (282.8)
Statistical Analysis 1: Comparison: Immune Naive vs Immune Resistant; Test type: Superiority; p = 0.71, Log Rank

ADVERSE EVENTS:
Time Frame: 36 months
Description: The study period during which adverse events must be reported is normally defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. For this study, the study treatment follow-up is defined as 30 days following the last administration of study treatment. Thereafter, only non-hematological related AEs of Grade 3 and can reasonably be attributed to the study treatment will be reported.
Arm/Group | Bone or Lung Index Lesion | Liver or Subcutaneous Index Lesion
All-Cause Mortality (participants affected / at risk) | 4/8 | 11/14
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/14
Other Adverse Events (participants affected / at risk) | 8/8 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bone or Lung Index Lesion (N=8) | Liver or Subcutaneous Index Lesion (N=14)
Atrial flutter and Shortness of Breath (Cardiac disorders) | 1 | 0 — This was a serious, expected AE that is not related to research and considered worsening of patient's heart disease.
Abdominal pain (Gastrointestinal disorders) | 0 | 1 — This is a serious, unexpected AE that is not related to research and is considered worsening of patient's disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bone or Lung Index Lesion (N=8) | Liver or Subcutaneous Index Lesion (N=14)
Colitis (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 6
Fatigue (General disorders) | 6 | 5
Fevers (General disorders) | 2 | 2
Chills (General disorders) | 2 | 1
Nausea (General disorders) | 3 | 2
Pain (General disorders) | 8 | 13
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Weight loss (Investigations) | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 1
Burning sensation at inguinal area (Reproductive system and breast disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dark/Blood urine (Renal and urinary disorders) | 1 | 1
Hemorroids (Gastrointestinal disorders) | 2 | 0
Hypophysitis (Endocrine disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lump in throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hypertension (Cardiac disorders) | 0 | 1
Hypercholesterolemia (Cardiac disorders) | 0 | 1
Insomnia (General disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hemianopsia (Eye disorders) | 0 | 3
Lump in right breast (Reproductive system and breast disorders) | 0 | 1
Worsening balance (General disorders) | 0 | 2
Lower jaw instability (Nervous system disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Bruising from fall (General disorders) | 1 | 0
Tingling in toes (General disorders) | 1 | 0
Edema (Lower extremities) (Vascular disorders) | 2 | 1
Anemia (Investigations) | 1 | 1
Hernia (Gastrointestinal disorders) | 1 | 0
Cancer sores (Skin and subcutaneous tissue disorders) | 0 | 1
Soft stool (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Numbness (Nervous system disorders) | 1 | 0
Weepy/teary (Psychiatric disorders) | 1 | 0
Cyst on left breast (Skin and subcutaneous tissue disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Swelling on right axillary region (General disorders) | 1 | 0
Stomach ache (Gastrointestinal disorders) | 1 | 2
Lightheadedness (Nervous system disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 1
Swelling in right neck (General disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Dysgeusia (General disorders) | 0 | 1
Cramps (Musculoskeletal and connective tissue disorders) | 1 | 1
Night sweats (General disorders) | 0 | 1
Hair loss (General disorders) | 0 | 1
Loss of appetite (Gastrointestinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Light sensitivity (General disorders) | 0 | 1
Tenderness/warmth of left neck (General disorders) | 0 | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Redness in axilla (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (General disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 0 | 1
Hemoptysis (General disorders) | 1 | 0
Altered mental status (Psychiatric disorders) | 1 | 0
Hypokalemia (Investigations) | 0 | 1
Leukocytosis (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
We stopped this trial early as the standard of care shifted during the course of the study. Participant flow, Baseline Characteristics and Adverse events were recorded as appropriate for the 23 patients (22 evaluable) who consented to the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT01970527/Prot_SAP_000.pdf